CLINICAL TRIAL: NCT03378609
Title: Prevalidation of the First German Version of the Vocal Fatigue Index (VFI)"
Brief Title: Prevalidation of the First German Version of the Vocal Fatigue Index (VFI)
Acronym: VFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: JB_2016-01511
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Vocal Fatigue
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vocal Fatigue Index (VFI) (Other): Standardized Questionnaire assessing vocal fatigue
  Interventions: Other: Vocal Fatigue Index (VFI)

INTERVENTIONS:
Other: Vocal Fatigue Index (VFI) — collection of 190 consecutive data sets, participants give separate consent for participating a retest or an interview, retest will be realised with the 10 following volunteers
  Other Names: Voice Handicap Index (VHI9i); Vocal Tract Discomfort Scale (VTD)

SUMMARY:
Vocal fatigue has been described as a common complaint in patients with voice disorders, however to date there is no standardized questionnaire in german language to assess specific symptoms. Main aim of this study is to assess the validity of the first german version of the Vocal Fatigue Index (VFI), and english questionnaire developed for voice patients to assess vocal fatigue.

In this study patients with voice disorders will receive the patient based questionnaires "Vocal Fatigue Index (VFI)", "Voice Handicap Index 9 international (VHI 9i)" and "Vocal Tract Discomfort Scale (VTD)", the study information and consent letter together with the standard invitation letter to a voice assessment at the Department for Phoniatrics and Speech Pathology University Hospital Zurich. Data of 93 consecutive volunteering patients will be collected. Furthermore a retest using the VFI will be conducted after 1 week with 10 volunteers. Thereafter construct validity of the VFI as compared to the established voice symptom questionnaires VHI 9i and VTD will be investigated. Further test-retest reliability will be determined.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* voice disorder (all etiologies)

Exclusion Criteria:

* age < 18 Jahre
* current voice therapy
* psychological disease
* botox injection in the Larynx
* inability to independently fill out the questionnaire

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Validity of the first German version ot the Vocal Fatigue Index (VFI) compared to the VHI9i and VTD | one day
  testing validity of the first German version ot the Vocal Fatigue Index (VFI) compared to the VHI9i and VTD

SECONDARY OUTCOMES:
Reliability of the first German version ot the Vocal Fatigue Index (VFI) compared to the VHI9i and VTD | one day
  testing reliability of the first German version ot the Vocal Fatigue Index (VFI) compared to the VHI9i and VTD

CONTACTS AND LOCATIONS:
Locations (1):
- ORL Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No